CLINICAL TRIAL: NCT03140059
Title: Comparison Between Surgical Access and Repeated Applications of APDT to Residual Pockets Treatment in Generalized Aggressive Periodontitis: Randomized Clinical Trial
Brief Title: Comparison Between Surgical Access and Repeated Applications of APDT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, DDS,MS,PhD, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SurgeryPDT
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Aggressive Periodontitis, Generalized
Keywords: surgical procedure; residual pockets; agressive periodontitis; antimicrobial photodynamic therapy
MeSH Terms: conditions — Aggressive Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open flap debridement (Active Comparator): In this group (n = 22), patients will receive open flap debridement will be performed to treat residual pockets.
  Interventions: Procedure: Open flap debridement
- Repeated application of aPDT (Active Comparator): In this group (n=22), patients will receive 5 applications of antimicrobial photodynamic therapy after the scaling and root planing.
  Interventions: Procedure: Repeated application of aPDT

INTERVENTIONS:
Procedure: Open flap debridement — Open flap debridement will be performed to decontaminate root surface
  Other Names: Surgical therapy
  Arms: Open flap debridement
Procedure: Repeated application of aPDT — Repeated application of photodynamic therapy (aPDT) at 0, 1, 2, 7 and 14 days post-operatively.
  Arms: Repeated application of aPDT

SUMMARY:
The aim of this study will be to compare the approach of repeated applications of APDT versus surgical therapy for the treatment of residual pockets in generalized agressive periodontitis.

DETAILED DESCRIPTION:
Scaling and root planing may be insufficient to resolve the periodontal infection resulting in residual periodontal pockets. A method of treatment to these sites would be the surgical therapy, because it allows access to root surfaces, making possible a better decontamination. However, the surgical approach may bring some negative points, as more discomfort and postoperative morbidity, increased transoperatory risk and increased risk of contamination. Thus, finding other alternatives to residual pockets treatment, antimicrobial photodynamic therapy (aPDT) was recently proposed. Therefore, the aim of this study will be to compare the approach of repeated applications of APDT versus surgical therapy for the treatment of residual pockets in generalized agressive periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of generalized aggressive periodontitis (Armitage, 1999; American Academy of Periodontology, 2015);
* Have undergone a first approach for periodontal treatment (full-mouth ultrasonic debridement);
* Present at least one residual pocket of probing depth ≥ 5 mm and bleeding on probe not located in furcation region;
* Good general health;
* Agree to participate in the study and sign the informed consent form (TCLE) after explaining the risks and benefits;

Exclusion Criteria:

* Systemic problems (cardiovascular alterations, blood dyscrasias, immunodeficiency - ASA III / IV / V) that contraindicate the periodontal procedure;
* Have used antibiotics and anti-inflammatories in the last six months;
* Smoke ≥ 10 cigarettes/day;
* Pregnant or lactating;
* Chronic use of medications that may alter the response of periodontal tissues;
* Indication of antibiotic prophylaxis for dental procedures;

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level | 6 months

SECONDARY OUTCOMES:
Probing depth | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, DDS, PhD, Study Director — Universidade Estadual Paulista "Julio de Mesquita Filho", ICT/UNESP

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lulic M, Leiggener Gorog I, Salvi GE, Ramseier CA, Mattheos N, Lang NP. One-year outcomes of repeated adjunctive photodynamic therapy during periodontal maintenance: a proof-of-principle randomized-controlled clinical trial. J Clin Periodontol. 2009 Aug;36(8):661-6. doi: 10.1111/j.1600-051X.2009.01432.x. Epub 2009 Jun 25. PMID 19563331